CLINICAL TRIAL: NCT04080466
Title: Cam Type Femoroacetabular Impingement (FAI) is a Cause of Hip Pain in the Young Adult and a Precursor to Osteoarthritis (OA)
Brief Title: Cam Type FAI is a Cause of Hip Pain in the Young Adult and a Precursor to OA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 20190456
Record Dates: First submitted 2019-08-22; First posted 2019-09-06 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Hip Dysplasia; Femoroacetabular Impingement; Osteoarthritis
Keywords: Hip; Cam deformity
MeSH Terms: conditions — Hip Dislocation; Femoracetabular Impingement; Osteoarthritis | interventions — Blood Specimen Collection; Urine Specimen Collection

STUDY DESIGN:
Intervention Model Description: Non-randomized, single centre trial with 2 parallel groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cam Group (Experimental): This group will consist of patients that are scheduled for surgery to undergo cam resection by hip arthroscopy.
  Interventions: Radiation: Low-dose CT Scan; Other: Blood/Urine Collection; Other: Patient Reported Questionnaires; Radiation: EOS Scan; Radiation: PET-MRI; Other: Motion Analysis; Radiation: 3T MRI
- Control Group (Active Comparator): This group will consist of a matched cohort of control participants.
  Interventions: Radiation: Low-dose CT Scan; Other: Blood/Urine Collection; Other: Patient Reported Questionnaires; Radiation: EOS Scan; Radiation: PET-MRI; Other: Motion Analysis; Radiation: 3T MRI

INTERVENTIONS:
Radiation: Low-dose CT Scan — Low dose computed tomography, also known as qCT, is sensitive to the mineral content within bone tissue, and can assess bone mineral density, a strong predictor of bone strength and stiffness, which can influence the health of the cartilage. Participants will undergo a low dose CT scan of both hips.
  Participants in the Cam Group will undergo this scan once as part of their standard of care. Participants in the Control Group will undergo this scan once as part of the study.
Other: Blood/Urine Collection — Collection of blood and urine allows the researchers to look for a biomarker in the blood and urine that might help to predict the evolution of disease/hip osteoarthritis. Identifying a marker in the blood and urine that could be used for early detection of individuals with cam deformity that are at-risk of hip degeneration could greatly improve patient care.
  Participants in the Cam Group will undergo the blood and urine collection twice; once before surgery and once 2-years post-operative. Participants in the Control Group will undergo a blood and urine collection once as part of the study.
Other: Patient Reported Questionnaires — The purpose of the questionnaires is to assess how much trouble the participant is having with their hip and how it affects their quality of life.
  Participants in the Cam Group will complete the questionnaires twice; once before surgery and once 2-years post-operative. Participants in the Control Group will complete the questionnaires once as part of the study.
Radiation: EOS Scan — The EOS® uses a new imaging technique that allows precise measurement of the hip and pelvis geometry and structure. This innovative x-ray technique exposes participants to 2-10 times less radiation than a routine x-ray and can capture multiple images at once.
  Participants in the Cam Group will undergo the EOS scan twice; once before surgery and once 2-years post-operative. Participants in the Control Group will undergo the scan once as part of the study.
Radiation: PET-MRI — Positron emission tomography combined with magnetic resonance imaging (PET-MRI) is a technology that allows physicians to examine bone and cartilage at the molecular level.
  Participants in the Cam Group will undergo the scan twice; once before surgery and once 2-years post-operative. Participants in the Control Group will undergo the scan once as part of the study.
Other: Motion Analysis — Motion analysis is the study of how joints move and which muscles fire during specific movements. In the lab, participants will be asked to perform movements that they might do during a typical day or when exercising.
  Participants in the Cam Group will undergo the Motion Analysis session twice; once before surgery and once 2-years post-operative. Participants in the Control Group will undergo the Motion Analysis session once as part of the study.
Radiation: 3T MRI — Participants will undergo a 3-Tesla (3T) Magnetic Resonance Imaging (MRI) of both hips.
  Participants in the Cam Group will undergo this scan once as part of their standard of care. Participants in the Control Group will undergo this scan once as part of the study.

SUMMARY:
An abnormally formed hip joint (cam deformity) is a major cause of osteoarthritis (OA). Individuals may not experience any symptoms until OA is severe due to extensive cartilage loss and changes in underlying bone. A series of studies showed that the cam deformity can lead to the development of OA if left untreated, thus strongly suggesting a causal relationship. Currently, the cam deformity that causes pain is surgically removed to relieve the pain and treat the associated cartilage damage. Recent studies have demonstrated that surgical treatment leads to bone and cartilage changes that were related to improved function and reduced pain.

DETAILED DESCRIPTION:
This study will allow the investigators to gain a better understanding of the relationship between cartilage and bone changes. The investigators will examine adult participants in the disease state that require surgical correction and compare to age-matched controls. The investigators will look at the impact of surgical intervention through joint-specific biomarkers of OA, specifically the PET-MRI and blood/urine biomarkers, which will allow them to simultaneously query cartilage and bone activity. The investigators propose that the use of PET-MRI will give more sensitive and hip-specific information about the joint health compared to the blood/urine biomarkers in patients with symptomatic cam morphology. Participants will undergo motion analysis and 3D modeling to help the investigators better understand the disease process during the performance of specific activities and define joint contact mechanics as they relate to the PET-MRI imaging, validating a biomarker for early joint degeneration. This diagnostic tool will be extremely useful for younger individuals with a cam deformity who have not yet developed symptoms. In the future the investigators could use this to detect early degeneration in adolescents to prevent and mitigate development of OA later on. This will also help the investigators develop activity guidelines for people with smaller cam deformities in order to avoid surgery and prevent degeneration.

ELIGIBILITY:
Inclusion Criteria:

* Skeletally mature patient undergoing cam resection by hip arthroscopy with hip pain longer than 6 months
* Absence of arthritis (Tonnis Grade 0 or 1)
* Absence of dysplasia (LCEA > 25°) or overcoverage (LCEA > 39°)
* Alpha angle greater than 55° on multiplanar imaging
* Subject is over the age of 18 years old at time of enrollment
* Subject is willing and able to complete required study visits and assessments
* Subject is willing to sign the approved Informed Consent Form

Group 2 Inclusion Criteria:

* Normal femoral head neck contour and no evidence of dysplasia
* Subject is over the age of 18 years old at time of enrollment
* Subject is willing and able to complete required study visits and assessments
* Subject is willing to sign the approved Informed Consent Form

Exclusion Criteria:

* Prior joint replacement surgery in any lower-limb joint due to OA
* History of lower-limb joint or back injury in the last year that impairs mobility
* Metallic prosthesis
* Worked with metal, metal fragments in the eye
* Blood transmittable disease(s)
* In vivo devices (Aneurysm clip(s), Pacemaker, ICD, Implanted hearing device)
* Extreme claustrophobia
* Overweight or obese (BMI > 30) and/or waist circumference >102cm in men and >88cm in women
* Diagnosis of Parkinson's or uncontrollable tremors
* Known history of early OA in the immediate family
* Pregnant, Breastfeeding, or planning to get pregnant
* Cognitive impairment that prevents accurate completion of patient-reported outcome questionnaires
* Patient unable/unwilling to complete all required follow-up visits
* Participants who have been exposed to other sources of radiation within the last year (Bringing radiation exposure above annual maximum)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2021-02-20 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of [18F]-NaF as a biomarker of hip degeneration | 24 months
  This study will assess [18F]-NaF uptake in PET-MRI as a novel biomarker of hip degeneration. This will be done by evaluating the presence of active bone turnover.

SECONDARY OUTCOMES:
Change in PET-MRI (SUV/T1Rho) | 24 months
  Determine the change in PET-MRI (SUV/T1Rho) two years after surgical correction of a symptomatic cam deformity to discern disease state.
qCT (Low Dose Computed Tomography) | Within 2 months after recruitment
  Used to measure bone mineral density (mass of mineral per volume of bone) in the subchondral bone. Negative scores indicate lower bone density, and positive scores indicate higher.
Change in type II collagen telopeptide (CTX-II) | 24 months
  Determine the change in urine biomarker levels (type II collagen telopeptide (CTX-II), measured by the ELISA kit, two years after surgical correction of a symptomatic cam deformity.
Change in cartilage oligomeric matrix protein (COMP) | 24 months
  Determine the change in serum biomarker levels (cartilage oligomeric matrix protein (COMP)), measured by the ELISA kit, two years after surgical correction of a symptomatic cam deformity.
Change in C-reactive protein (CRP) | 24 months
  Determine the change in serum biomarker levels (C-reactive protein (CRP)), measured by the ELISA kit, two years after surgical correction of a symptomatic cam deformity.
Change in N-terminal cross-linking telopeptide of type I collagen (NTX-1) | 24 months
  Determine the change in bone turnover plasma biomarker levels (N-terminal cross-linking telopeptide of type I collagen (NTX-1)) two years after surgical correction of a symptomatic cam deformity.
Change in carboxy-terminal collagen crosslinks (CTx) | 24 months
  Determine the change in bone turnover plasma biomarker levels (carboxy-terminal collagen crosslinks (CTx)), measured by the ELISA kit, two years after surgical correction of a symptomatic cam deformity.
Change in N-terminal pro-peptide of type I procollagen (PINP) | 24 months
  Determine the change in bone turnover serum biomarker levels (N-terminal pro-peptide of type I procollagen (PINP)), measured by the ELISA kit, two years after surgical correction of a symptomatic cam deformity.
Change in iHot-33 score | 24 months
  The International Hip Outcome Tool (iHOT-33 is a questionnaire that evaluates young active patients with early hip disease. The questionnaire is self-administered and assesses across 4 domains: symptoms and functional limitations; sport and recreational activities; job-related concerns; and social, emotional, and lifestyle concerns. Questions are answered by marking a visual analog scale between 2 anchor statements (100-mm scale). The total score is calculated as a simple mean of these responses ranging from 0 to 100, with 100 representing the best possible quality-of-life score.
Change in Hip Disability and Osteoarthritis Outcome Score (HOOS) score | 24 months
  Hip-specific symptoms and functional impairment will be compared using the Hip Disability and Osteoarthritis Outcome Score (HOOS). This 40-item patient reported outcome tool has 5 categories: pain, symptoms, daily living, quality of life, sports and recreational activities. Each category is scored on 100 points, 0 being the worse outcome and 100 the best outcome.
Change in EQ-5D-5L score | 24 months
  This questionnaire assesses generic health status. Each question is scored from 1-5, with 1 being no problems and 5 being severe problems. These scores are not aggregated. There are 5 domains: mobility, self-care, usual activities, pain and anxiety. The final question is asking the participant to self score their health that day out of 100 (0 being the worst health and 100 being the best health).
Joint Kinematics to predict hip contact forces | 24 months
  Retro-reflective markers will be placed on each participant in a laboratory setting. Joint kinematics will be reconstructed from marker trajectories recorded by a 10- camera system (Vicon Vantage & Vicon Vero, Oxford, UK; frequency 200 Hz). Together, with joint kinetics, the investigators will predict hip contact forces.
Joint kinetics to predict hip contact forces | 24 months
  Retro-reflective markers will be placed on each participant in a laboratory setting. Force platforms will record kinetic data. Together, with joint kinetics, the investigators will predict hip contact forces.
Muscle Activity | 24 months
  Retro-reflective markers will be placed on each participant in a laboratory setting. Electromyography (EMG) electrodes will be placed over the following muscles: rectus femoris, vastus medialis, vastus lateralis, tensor fascia latea, biceps femoris, semitendinosus, gluteus medius and gluteus maximus. Muscle activity will be measured using EMG signal recorded during maximum voluntary isometric contraction.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Beaule, MD, FRCSC, Principal Investigator — The Ottawa Hospital Research Institute
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No